CLINICAL TRIAL: NCT00329498
Title: Manipulation of L-Ascorbic Acid Level For The Treatment of Selected Cases Of Acute Myeloid Leukemia and Myelodysplastic Syndromes
Brief Title: L-Ascorbic Acid Depletion to Treat Acute Myeloid Leukemia and Myelodysplastic Syndromes
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Jin Yang Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMCIRB-98-04-02
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: ascorbic acid
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Ascorbic Acid

INTERVENTIONS:
Drug: L-Ascorbic Acid

SUMMARY:
To document therapeutic gain achieved by cyclic application of L-ascorbic acid (LAA) supplementation and depletion, while confirming safety and avoidance of clinically significant scurvy, in chemorefractory patients with acute myeloid leukemia (AML) and myelodysplastic syndromes (MDS).

DETAILED DESCRIPTION:
The seminal discovery that the in vitro growth of malignant cells could be absolutely dependent on L-ascorbic acid (LAA) was originally published in Sciene. The cell culture assay used with a mouse plasmacytoma model in this discovery was based on colony formation, and was essentially the same as the one used to grow normal hemopoietic colonies, such as CFU-GM and CFU-G, from normal bone marrow specimens. Subsequent analysis of the growth factors for these CFUs using this same culture system eventually led to the discovery of colony stimulating factors, such as GM-CSF and G-CSF, now widely used clinically. Human leukemia, specifically acute myeloid leukemia (AML), cell colonies also grow well in this culture system, as shown by extensive cell biology studies. In addition, cells from patients with myelodysplastic syndrome (MDS), a significant proportion of them progressing to AML behave similarly to AML cells in this culture system . In particular both AML and MDS are identical in that the growth of colonies is enhanced by addition of LAA to the cell culture media in a high proportion of these patients.

The large volume of in vitro data thus generated, including correlations with direct clinical relevance is increasingly convincing that lowering of LAA levels could potentially be developed and utilized as a treatment for specific hemopoeitic malignancies. This was particularly attractive in view of the fact that the growth of normal hemopoietic colonies, such as CFU-GM and CFU-G, is never enhanced by LAA. Such an absolute selectivity would predict a lack of clinical adverse hemopoetic events from an intervention which lowered LAA levels. We also had seemingly-contradictory data that the growth of colonies from AML and MDS patients could be suppressed by addition of LAA, infrequently but sometimes profoundly. However, detailed dose response analysis later clarified this: low physiologic doses enhance and high pharmacologic doses suppress formation of leukemic colonies. From a therapeutic perspective, we would have greater expectations for a depletion strategy than for supplementation, because 1) leukemic suppression by addition of LAA is often accompanied by some mild suppression of the normal CFU and therefore is not absolutely selective; and 2) LAA supplementation has been clinically tested in a variety of solid tumors, with controversial outcomes.

Therefore, our original protocol was developed primarily to accomplish lowering of LAA levels, with a subsequent oral LAA supplementation used primarily to prevent scurvy and only secondarily for possible benefit. However, with the first patient there was a strong indication of antileukemic effects during both the LAA depletion and supplementation phases. Based on this encouragement, the protocol was amended to formally alternate depletion with supplementation, and to utilize intravenous (IV) administration of LAA to achieve high dose supplementation. With 17 subsequent subjects having been treated, this study of the safety and efficacy of cyclic manipulation of LAA levels has demonstrated beneficial outcome in a high proportion of refractory and terminal patients with AML or MDS. Moreover, growing laboratory evidence being produced provides a molecular basis for these clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have AML or MDS according to new WHO classification, with minimum of 5% blasts in peripheral blood.
* There must be a clear and acceptable reason for not receiving standard treatments (chemotherapy and/or stem cell transplantation); or standard treatments have already been given and this option exhausted with evidence of refractory disease.
* Prior treatments of any forms are allowed provided there is no potential residual beneficial effect and the patients are off treatment for at least 4 weeks, with estimated life expectancy of at least 2 months.
* Adequate amount (4 ml) of bone marrow sent to the laboratory for cell culture studies.
* There are no restrictions based on age, sex, or ethnicity except that adequate contraception must be practiced in women of childbearing ages. Although AML is rare in children, pediatric patients will be accepted.
* There is no deficiency of G6PD (RBC).
* Asymptomatic patients with disease progression and symptomatic patients.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1998-05; Study Completion 2005-08

PRIMARY OUTCOMES:
Efficacy
Safety, clinically

SECONDARY OUTCOMES:
Correlative studies between the modulation of the growth of leukemic colony-forming-cells(CFC) by L-ascorbic acid (LAA) in cell-culture and clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Park CH, Kimler BF, Yi SY, Park SH, Kim K, Jung CW, Kim SH, Lee ER, Rha M, Kim S, Park MH, Lee SJ, Park HK, Lee MH, Yoon SS, Min YH, Kim BS, Kim JA, Kim WS. Depletion of L-ascorbic acid alternating with its supplementation in the treatment of patients with acute myeloid leukemia or myelodysplastic syndromes. Eur J Haematol. 2009 Aug;83(2):108-18. doi: 10.1111/j.1600-0609.2009.01252.x. Epub 2009 Mar 5. PMID 19284416